CLINICAL TRIAL: NCT05565235
Title: Efficacy of Serratus Anterior Plane Block Using Bupivacaine Alone, Bupivacaine/ Magnesium Sulfate Versus Bupivacaine/ Nalbuphine for Thoracotomy: A Randomized, Double-Blinded Comparative Study.
Brief Title: Comparing Efficacy of Different Drugs Combinations for Serratus Anterior Block for Thoracotomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hussein Sayed Hasan, lecturer of anesthesia , surgical ICU and pin managment, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: N-50-2022
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Post Operative Pain, Acute
Keywords: thoracotomy; serratus anterior plane block
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Magnesium; Nalbuphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: patient doesn't know which type of drugs given to him in the block , and the investigator who collect postoperative data also doesn't know which type of drugs used in the block
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group B (Active Comparator): bupivacaine
  Interventions: Drug: patients will receive intraoperative serratus block with bupivacaine
- Group BMG (Active Comparator): bupivacaine/ magnesium.
  Interventions: Drug: serratus block with bupivacaine /magnesium
- Group BN (Active Comparator): bupivacaine /nalbuphine.
  Interventions: Drug: serratus block with bupivacaine with nalbuphine

INTERVENTIONS:
Drug: patients will receive intraoperative serratus block with bupivacaine — no additives
  Arms: Group B
Drug: serratus block with bupivacaine /magnesium — magnesium added
  Arms: Group BMG
Drug: serratus block with bupivacaine with nalbuphine — nalbuphine added
  Arms: Group BN

SUMMARY:
We aim to compare efficacy and efficiency of serratus anterior block with bupivacaine alone to bupivacaine/magnesium and bupivacaine /nalbuphine in postoperative analgesia for thoracotomy surgery.

Objectives:

To compare bupivacaine alone, bupivacaine/magnesium and bupivacaine /nalbuphine in serratus anterior plane block for intraoperative and postoperative analgesia for thoracotomy surgery.

* The time for 1st rescue analgesia.
* Calculation of the opioid requirements; (the total intra-operative post-operative morphine consumption in first 24h postoperative).
* Assessment of pain score (VAS)- rest, VAS-movement, VAS-cough during post-operative 24hrs period.

Hypothesis:

We hypothesize that magnesium sulfate and nalbuphine can reduce acute postoperative pain and result in efficacious postoperative analgesia due to block of the lateral cutaneous branches of the intercostal nerves (T2 - T6) by diffusion across the inter-fascial planes.

DETAILED DESCRIPTION:
I. Study design prospective, randomized controlled study. II. Study setting and location It will be conducted at El Kasr Al-Aini hospitals, cardiothoracic Surgery, Cairo University.after registration in clinicaltrials.gov and getting a unique number III. Study population patients of both genders, aged (16 - 65) years old, ASA I, II or III scheduled for elective general thoracotomy surgeries will be included. Consenting patients will be randomly allocated to one of three groups: Group B: patients will receive intraoperative serratus block with bupivacaine. Group BMG: patients will receive intraoperative serratus block with bupivacaine/ magnesium.

Group BN: patients will receive intraoperative serratus block with bupivacaine /nalbuphine.

V. Study Procedures

1. Randomization:

   The patients will be randomized using a computer-generated list of random numbers which will be sealed in closed envelopes. Patients will be randomly allocated to one of the three groups. The study drugs are going to be prepared by anesthetist (who were blinded to the study and did not share in the technique) in labelled syringes, patients into 3 groups by a sealed opaque envelope, and received the study drug as follows: group B (n = 26): (bupivacaine): received bupivacaine 30 mL 0.25%, group BMG (n =26): received bupivacaine 30 mL 0.25% and 500 mg magnesium sulphate. Group BN (n =26): (bupivacaine/nalbuphine): received bupivacaine 30 mL 0.25 % and nalbuphine 0.2 mg/kg.
2. Study Protocol All patients will be assessed clinically and investigated for exclusion of any of the above-mentioned contraindications.

Laboratory work needed will be: Complete blood count (CBC); prothrombin time and concentration (PT& PC, INR), renal functions and liver function tests or other necessary investigation for the desired surgery. ECG, CXR, CT chest and echocardiography will be done if needed preoperatively Anesthetic application

* Standard monitoring procedures will include continuous ECG, pulse oximetry, invasive arterial blood pressure, end-tidal CO2, inhaled gas analyzer and temperature monitoring. Baseline readings (T0) of heart rate, systolic, diastolic, and mean blood pressure are going to be record after monitor attachment and every 30 min
* General anesthesia will be induced in all groups (B, BN, AND BMG group) using fentanyl 2 mic/kg, propofol 2 mg/kg and atracurium 0.5 mg/kg while in obese patients Lean body weight (LBW) will be used. single or double lumen tube will be used as preferred by surgeon, Anesthesia will be maintained using isoflurane (1 MAC) and atracurium supplements were given to maintain muscle relaxation., diclofenac 75mg once iv infusion and acetaminophen 15 mg/kg. Additional dose of fentanyl 1mic / kg will be given if there is tachycardia >100 or intraoperative hypertension more than 20% of the preoperative value. In addition to, all patients will receive cefotaxime 50 mg/kg.

Near the end of surgery, the surgeon is going to aspirate the content of the labelled syringes with a sterile one and ask to inject it below the serratus anterior muscle after closing it. To prevent inadvertent intravascular insertion of the needle, the study drugs are going to be injected in increments after repeated aspiration. At the end of the surgery, inhaled anesthetic is going to discontinue. After the reversal of muscle relaxation and full recovery, patients will be monitored at the recovery unit. Postoperative pain Visual Analogues Scales (VAS, VAS movement, VAS cough) are going to be measure pain (static, dynamic and with cough respectively), where 0 = "no pain" and 10 = "worst pain imaginable", at 1, 6, 12, 24 h by a person not oriented by protocol. Classic postoperative analgesic regimen (Diclofenac 75mg every 8hrs and acetaminophen 1gm every 6 hrs.). The efficacy of the block will be test by measuring the distribution of lost cold sensation along distribution of lateral cutaneous nerve from second intercostal to ninth intercostal nerve.

Morphine 2 mg Iv incremental boluses will be given as rescue analgesia for patients if VAS score >3.

1. Measurement tools

* Demographic data (age, sex, BW) patient surgery characteristic (duration of the surgery, type of operation) and ASA status will be recorded.
* In the PACU and the ward, patient will be assessed for the first 24 hours post-operative period using (VAS score) for Pain assessment.

Blood pressure (SBP, DBP and MAP) and heart rate will also be recorded during the operation and the first 24 hours post-operative period and intraoperative fentanyl doses.

Statistical Analysis I. Sample size The time of 1st use of rescue analgesia post-operatively is defined as the primary outcome of the study using one-way ANOVA test. As based on previous study (Comparison of ultrasound-guided serratus plane block and thoracic paravertebral block for postoperative analgesia after thoracotomy, a randomized controlled trial Research and Opinion in Anesthesia & Intensive Care 2018, 5:314-322), the mean time to 1st use of morphine was (6.2 ± 1.66) hours.

If combining the bupivacaine with nalbuphine or with magnesium would result in a 30% increase in the time to 1st use of morphine: α error of 0.05 and power of 0.95. A minimum of 78 patients was calculated (27 patients in each group). sample size was calculated using G-Power version 3.1.9.2 software.

II. Statistical analysis

Analysis of data will be performed using Statistical package for social science (SPSS) software, version 15 for Microsoft Windows (SPSS Inc., Chicago, IL, and USA). Categorical data will be reported as numbers and percentages and will be analyzed using chi-squared test. Continuous data will be checked for normality using Kolmogorov-Smirnov test. Normally distributed data will be presented as means (standard deviations) and will be analyzed using unpaired student t-test. Skewed data will be expressed as medians (quartiles) and will be analyzed using Mann Whitney U test. For repeated measures, a two-way repeated measure ANOVA will be used to evaluate the block (between-groups factor) and the time (repeated measures)". Post-hoc pairwise comparison will be performed using Bonferroni test. P value of 0.05 or less will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Elective thoracotomy or unplanned thoracotomy after failed thoracoscopic surgery
* Patient with American Society of Anesthesiology ASA I, II or III.

Exclusion Criteria:

1. Patient refusal
2. Contraindication for regional anesthesia

   * Allergy from local anesthetics
   * Bleeding diathesis (Bleeding tendency with prothrombin concentration PC less than 75 % or platelet count less than 50,000/µL.
   * Use of anticoagulants, infection at the puncture site.
3. Presence of severe Chronic renal impairment or acute renal failure, decompensated liver disease, cardiac or psychiatric disorders, GIT ulcers, communication barriers, hearing deficit or high grades of visual deficit that interfere with consenting, VAS assessments, and delirium, or another cognitive dysfunction.
4. Patient intubated preoperatively.
5. Patient will not be extubated immediately postoperatively
6. Opioid tolerant patients.
7. Any contraindications of Magnesium infusion as hypovolemia or severe impaired ventricular systolic function.
8. Contraindication of acetaminophen and Diclofenac sodium administration.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-12-09 (Actual); Primary Completion 2023-09-10 (Estimated); Study Completion 2023-11-10 (Estimated)

PRIMARY OUTCOMES:
The time of 1st rescue analgesia post operative | one year
  if VAS or VAS-movement >3.

SECONDARY OUTCOMES:
Pain assessment score; (VAS score) VAS-movement and VAS-cough | one year
  at 1, 6, 12, 24 hours post-operative period
Total amount of morphine (mg) used in 24h post operatively | one year
  when VAS >3
Hemodynamic changes (SBP, DB, MAP) | one year
  during the first 24 hours in the postoperative period
Incidence of local anesthetic toxicity. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Tamer M. Atteya, M.D, Study Chair — Lecturer of anesthesia,surgical ICU and pain managment
Locations (1):
- Kasr Alainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gerner P. Postthoracotomy pain management problems. Anesthesiol Clin. 2008 Jun;26(2):355-67, vii. doi: 10.1016/j.anclin.2008.01.007. PMID 18456219
- [Background] Kavanagh BP, Katz J, Sandler AN. Pain control after thoracic surgery. A review of current techniques. Anesthesiology. 1994 Sep;81(3):737-59. doi: 10.1097/00000542-199409000-00028. No abstract available. PMID 8092520
- [Background] Katz J, Jackson M, Kavanagh BP, Sandler AN. Acute pain after thoracic surgery predicts long-term post-thoracotomy pain. Clin J Pain. 1996 Mar;12(1):50-5. doi: 10.1097/00002508-199603000-00009. PMID 8722735
- [Background] Kaushal B, Chauhan S, Saini K, Bhoi D, Bisoi AK, Sangdup T, Khan MA. Comparison of the Efficacy of Ultrasound-Guided Serratus Anterior Plane Block, Pectoral Nerves II Block, and Intercostal Nerve Block for the Management of Postoperative Thoracotomy Pain After Pediatric Cardiac Surgery. J Cardiothorac Vasc Anesth. 2019 Feb;33(2):418-425. doi: 10.1053/j.jvca.2018.08.209. Epub 2018 Aug 31. PMID 30293833
- [Background] Semyonov M, Fedorina E, Grinshpun J, Dubilet M, Refaely Y, Ruderman L, Koyfman L, Friger M, Zlotnik A, Klein M, Brotfain E. Ultrasound-guided serratus anterior plane block for analgesia after thoracic surgery. J Pain Res. 2019 Mar 11;12:953-960. doi: 10.2147/JPR.S191263. eCollection 2019. PMID 30881105
- [Background] De Oliveira GS Jr, Castro-Alves LJ, Khan JH, McCarthy RJ. Perioperative systemic magnesium to minimize postoperative pain: a meta-analysis of randomized controlled trials. Anesthesiology. 2013 Jul;119(1):178-90. doi: 10.1097/ALN.0b013e318297630d. PMID 23669270
- [Background] Chawda PM, Pareek MK, Mehta KD. Effect of nalbuphine on haemodynamic response to orotracheal intubation. J Anaesthesiol Clin Pharmacol. 2010 Oct;26(4):458-60. PMID 21547169